CLINICAL TRIAL: NCT01262677
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group, Multi-center Trial Of Pregabalin Controlled Release Formulation As Adjunctive Therapy In Adults With Partial Onset Seizures
Brief Title: Once-A-Day Pregabalin For Partial Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A0081194; 2010-019035-35 (EudraCT Number)
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2018-04

CONDITIONS: Partial Seizures; Epilepsies, Partial
Keywords: Partial epilepsy; partial seizures; epilepsy; seizures; adjunctive therapy; intervention; controlled-release; placebo-controlled; seizure
MeSH Terms: conditions — Seizures; Epilepsies, Partial; Epilepsy | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- pregabalin CR 330 mg (Experimental)
  Interventions: Drug: pregabalin
- pregabalin CR 165 mg (Experimental)
  Interventions: Drug: pregabalin
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pregabalin — Controlled Release Tablets, 82.5 mg, once per day (QD) for 3 days
  Arms: pregabalin CR 330 mg
Drug: pregabalin — Controlled Release Tablets, 165 mg, once per day (QD) for 11 days
  Arms: pregabalin CR 330 mg
Drug: pregabalin — Controlled Release Tablets, 330 mg, once per day (QD) for the remainder of the double-blind treatment phase (max is 12 weeks)
  Arms: pregabalin CR 330 mg
Drug: pregabalin — Controlled Release Tablets, 165 mg, once per day (QD) for 7 days
  Arms: pregabalin CR 330 mg
Drug: pregabalin — Controlled Release Tablets, 82.5 mg, once per day (QD) for 3 days
  Arms: pregabalin CR 165 mg
Drug: pregabalin — Controlled Release Tablets, 165 mg, once per day (QD) for the remainder of the up-titration and double-blind treatment and taper phases (max 14.5 weeks)
  Arms: pregabalin CR 165 mg
Drug: placebo — matched to the active drug
  Arms: Placebo

SUMMARY:
Approximately 30% percent of subjects with partial seizures are refractory to treatment with single or combination antiepileptic drugs. The present study will compare the efficacy of two different dosages of pregabalin CR dosed once daily as compared to placebo, when used as adjunctive therapy in subjects requiring adjunctive therapy for partial onset epilepsy, using a randomized, parallel group design.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of epilepsy with partial onset seizures (seizures may be simple or complex, with or without evolution into a bilateral, convulsive seizure)
* Currently taking 1 to 3 anti-epilepsy medicines (AEDs) at stable dosages, and who have taken at least 2 prior (or ongoing) AEDs

Exclusion Criteria:

* Primary generalized seizures (for example, absence, myoclonic seizures or Lennox-Gastaut Syndrome)
* Status epilepticus within one year prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2011-02-17 (Actual); Primary Completion 2012-07-31 (Actual); Study Completion 2012-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (82):
- United States (26):
  - Neurology Clinic, PC, Northport, Alabama
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - Clinical Trials, Inc., Little Rock, Arkansas
  - Collaborative Neuroscience Network, Inc., Long Beach, California
  - Viking Clinic Research Center, Murrieta, California
  - Viking Clinical Research Center, Murrieta, California
  - Neurological Research Institute, Santa Monica, California
  - Viking Clinical Research Center, Temecula, California
  - Sarkis Clinical Trials, Gainesville, Florida
  - Optima Neurological Services, LLC, Gainesville, Florida
  - Sleep Disorders Center of Georgia - Gainesville, Gainesville, Georgia
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - VCMA Comprehensive Epilepsy Center, Wichita, Kansas
  - Via Christi Research, Wichita, Kansas
  - Associates in Neurology, PSC, Lexington, Kentucky
  - Mid Atlantic Headache Institute, Pikesville, Maryland
  - Asheville Neurology Specialists, PA, Asheville, North Carolina
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Mark A. Fisher, M.D.- Private Practice, Oklahoma City, Oklahoma
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Veroniqe Sebastian, MD, Oklahoma City, Oklahoma
  - Angelique Barreto, MD, Oklahoma City, Oklahoma
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - FutureSearch Trials of Neurology, Austin, Texas
  - Scott and White Healthcare-Office of Sponsored Research Administration, Temple, Texas
  - Scott & White Healthcare, Temple, Texas
- Fundacion Argentina Contra las Enfermedades Neurologicas (FACENE), Buenos Aires, Argentina
- Clinic of Neurology,Clinical Centar University Sarajevo, Sarajevo, Bosnia and Herzegovina
- Bulgaria (5):
  - MBAL Puls AD, Nevrologichno otdelenie, Blagoevgrad
  - UMBAL Dr. Georgi Stranski, Vtora nevrologichna klinika, Pleven
  - DKTs Akta Medika, Konsultativen kabinet po Nevrologiya, Sevlievo
  - MBALNP Sveti Naum EAD, Klinika po nervni bolesti za paroksizmalnite sastoyaniya,, Sofia
  - Vtora Mnogoprofilna Bolnitsa za Aktivno Lechenie, Nevrologichno Otdelenie, Sofia
- Czechia (3):
  - Litomyslská nemocnice, a.s., Litomyšl
  - Fakultni Thomayerova nemocnice s poliklinikou,Neurologicka klinika IPVZ/FTNsP, Prague
  - Neurologicka ambulance, Prague
- Germany (6):
  - Epilepsie-Zentrum Bethel, Bielefeld
  - Praxis fuer Neurologie und Psychiatrie, Psychotherapie, Bielefeld
  - Klinik fuer Epileptologie, Universitaet Bonn, Bonn
  - Neuro Consil GmbH, Düsseldorf
  - Epilepsieklinik fuer Erwachsene Epilepsiezentrum Kork, Kehl-Kork
  - Studienzentrum Dr. Stephan Arnold, München
- Hong Kong (2):
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Department of Medicine, Queen Elizabeth Hospital, Kowloon
- Hungary (4):
  - Dr. Kennessey Albert Korhaz-Rendelointezet, Neurologiai Osztaly, Balassagyarmat
  - Synexus Magyarorszag Kft., Budapest
  - Fovarosi Onkormanyzat Uzsoki utcai Korhaza, Ideggyogyaszati Osztaly, Budapest
  - Szent Pantaleon Korhaz Nonprofit Kft., Idegosztaly, Dunaújváros
- India (8):
  - Lalitha Super Specialities Hospital (P) Ltd., Guntur, Andhra Pradesh
  - Jagadguru Sri Shivathreeshwara Medical College and Hospital,, Mysore, Karnataka
  - Deenanath Mangeshkar Hospital and Research Centre, Pune, Maharashtra
  - Sahyadri Clinical Research & Development Center,, Pune, Maharashtra
  - KEM Hospital Research Centre, Pune, Maharashtra
  - Sahyadri Speciality Hospital, Pune, Maharashtra
  - Poona Hospital and Research Centre Department of Neurology, Pune, Maharashtra
  - Vidyasagar Institute of Mental Health , Neuro& Allied Sciences,, Nehru Nagar, NEW Delhi
- Malaysia (3):
  - Jabatan Neurosains, Pusat Pengajian Sains Perubatan, Universiti Sains Malaysia., Kubang Kerian, Kelantan
  - Hospital Universiti Sains Malaysia, Kelantan Darul Naim
  - Hospital Kuala Lumpur, Kuala Lumpur
- Mexico (5):
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara, Jalisco
  - Private Office 201, Delagación Cuauhtemoc, Mexico City
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Hospital Angeles Culiacan, Culiacán, Sinaloa
  - Instituto Biomedico de Investigacion A. C., Aguascalientes
- Poland (4):
  - Indywidualna Specjalistyczna Praktyka Lekarska, Gdansk
  - Centrum Neurologii Klinicznej Sp. z o. o., Krakow
  - Gabinet Lekarski A. Klimek, Lodz
  - Niepubliczny Zaklad Opieki Zdrowotnej IGNIS dr med. Alicja Lobinska, Świdnik
- Epilepsy Control Institute, San Juan, PR, Puerto Rico
- Romania (2):
  - Spitalul Clinic de Urgenta "Prof. Dr. Nicolae Oblu", Iași, JUD. IASI
  - Cabinet Medical Individual " Dr. Adina Maria Roceanu", Bucharest
- Russia (6):
  - Municipal Healthcare Institution City Hospital #5, Neurology Department, Barnaul
  - State Medical Institution Republican Clinical Hospital, Kazan'
  - Central Clinical Hospital #2 N.A. Semashko OAO RZD / Department of Rehabilitation, Moscow
  - Pyatigorsk City Hospital #2, Neurology Department,, Pyatigorsk
  - State Institution St. Petersburg Psychoneurological Research Institute V.M. Bekhterev of Roszdrav, Saint Petersburg
  - Samara Regional Clinical Hospital M.I. Kalinin, Neurology and Neurosurgery Department, Samara
- Institute for Mental Health, Belgrade, Serbia
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
- Thailand (2):
  - Khon Kaen University, Faculty of Medicine, Neurology Unit, Department of Medicine, Muang, Changwat Khon Kaen
  - Neurology Division, Department of Medicine, Pramongkutklao College of Medicine, Bangkok

REFERENCES:
- [Derived] French J, Brandt C, Friedman D, Biton V, Knapp L, Pitman V, Chew M, Dubrava S, Posner HB. Adjunctive use of controlled-release pregabalin in adults with treatment-resistant partial seizures: a double-blind, randomized, placebo-controlled trial. Epilepsia. 2014 Aug;55(8):1220-8. doi: 10.1111/epi.12690. Epub 2014 Jun 24. PMID 24962242
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081194&StudyName=Once-A-Day%20Pregabalin%20For%20Partial%20Seizures

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter, multinational study and included four standard phases: an 8-week baseline observation phase, a 2-week dose escalation phase, a 12-week fixed-dose maintenance phase, and a 1-week taper phase.
Pre-assignment Details: An 8-week baseline observation phase began immediately after the screening visit. Througout the observation phase the participants continued their current anti-epileptic drugs (AEDs) at the prescribed dosage, eligibility was re-evaluated at Week -4 and Week 0, and the participants recorded all seizures in daily seizure diaries.
Groups:
- Pregabalin 165 mg: After the 2-week dose escalation phase, the participants received 165 mg of pregabalin once a day during the 12-week double-blind maintenance phase. Afterwards, the study medication was tapered for one week. The tablets were to be taken orally, within 1 hour (hr) after the evening meal. The medication must have been taken intact and not bitten, chewed, cut, or otherwise altered prior to swallowing.
- Pregabalin 330 mg: After the 2-week dose escalation phase, the participants received 330 mg of pregabalin once a day during the 12-week double-blind maintenance phase. Afterwards, the study medication was tapered for one week. The tablets were to be taken orally, within 1 hr after the evening meal. The medication must have been taken intact and not bitten, chewed, cut, or otherwise altered prior to swallowing.
- Placebo: After the 2-week dose escalation phase, the participants received placebo once a day during the 12-week double-blind maintenance phase. Afterwards, the study medication was tapered for one week. The tablets were to be taken orally, within 1 hr after the evening meal. The medication must have been taken intact and not bitten, chewed, cut, or otherwise altered prior to swallowing.
Period: Overall Study
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Started | 100 | 113 | 110
Completed | 91 | 98 | 98
Not Completed | 9 | 15 | 12
Not completed — Does not meet entrance criteria | 0 | 2 | 0
Not completed — Insufficient clinical response | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 0 | 2
Not completed — No longer willing to participate | 3 | 3 | 2
Not completed — Reason not provided | 2 | 1 | 3
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Adverse Event (AE) related to study drug | 3 | 8 | 3

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all randomized participants who took at least one dose of the study medication.
Groups:
- Pregabalin 165 mg: After the 2-week dose escalation phase, the participants received 165 mg of pregabalin once a day during the 12-week double-blind maintenance phase. Afterwards, the study medication was tapered for one week. The tablets were to be taken orally, within 1 hr after the evening meal. The medication must have been taken intact and not bitten, chewed, cut, or otherwise altered prior to swallowing.
- Total: Total of all reporting groups
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo | Total
Number analyzed (Participants) | 100 | 113 | 110 | 323
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.88 (13.10) | 39.58 (13.15) | 38.72 (13.25) | 38.76 (13.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 55 | 61 | 169
  Male | 47 | 58 | 49 | 154

OUTCOME MEASURES:

1. Primary Outcome: Log Transformed (Loge) 28-day Seizure Rate for All Partial Onset Seizures During the Double-blind Treatment Phase
Description: Seizures were recorded and documented in a daily Seizure Diary by the participants, family member, caregiver, or legal guardian. Simple partial seizures without a visible motor component (ie, lacking visible movements during the seizure) were not counted toward eligibility, or in the primary or secondary efficacy analyses. Natural logarithm of the 28-day seizure rate was reported in this outcome measure.
Time Frame: Week 0 to Week 14
Population: The intent-to treat (ITT) population consisted of all randomized participants who received at least one dose of double-blind treatment, and had a baseline and at least one follow-up double-blind treatment phase assessment visit. The ITT population was the primary sample and included: Pregabalin 165 mg: 100, Pregabalin 330 mg: 112, Placebo: 109.
Measure: Mean (Standard Deviation); unit: ln (seizures per 28 days)
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 100 | 112 | 109
ln (seizures per 28 days)
  Baseline | 2.24 (0.757) | 2.33 (0.873) | 2.32 (0.910)
  Week 14: number analyzed (Participants) | 98 | 111 | 109
  Week 14 | 1.84 (1.003) | 1.80 (1.030) | 1.93 (1.132)
Statistical Analysis 1: Comparison: Pregabalin 165 mg vs Placebo; ANCOVA model with the following fixed terms was used to calculate the p-value: loge (baseline 28-day seizure rate + 1) as a coninuous covariate, sites pooled by geographic region (ie, U.S., Europe, Asia, rest of the world), and treatment group (placebo, pregabalin 165 mg controlled-release (CR), pregabalin 330 mg CR). 88 participants in each group (264 total) should have provided approximately 90% power; Test type: Superiority; p = 0.9076, ANCOVA — Statistical testing was done at 95% confidence intervals, two-sided, least square means and their standard errors; Mean Difference = -0.99, 95% CI 2-sided [-16.28 to 17.11] — Value is percent reduction in seizures relative to placebo
Statistical Analysis 2: Comparison: Pregabalin 330 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0907, ANCOVA — Statistical testing was done at 95% confidence intervals, two-sided, least square means and their standard errors; Mean Difference = -13.05, 95% CI 2-sided [-26.07 to 2.25] — Value is percent reduction in seizures relative to placebo

2. Secondary Outcome: Percentage of Participants With a ≥50% Reduction in the 28-day Partial Seizure Rate From Baseline During the Double-blind Treatment Phase
Description: Seizures were recorded and documented in a daily Seizure Diary by the participants, family member, caregiver, or legal guardian. Simple partial seizures without a visible motor component (ie, lacking visible movements during the seizure) were not counted toward eligibility, or in the primary or secondary efficacy analyses. Participants who had a ≥50% reduction in the 28-day partial seizure rate from baseline were defined as a responder, otherwise they were default as a non-responder.
Time Frame: Week 0 to Week 14
Population: The ITT population consisted of all randomized participants who received at least one dose of double-blind treatment, and had a baseline and at least one follow-up double-blind treatment phase assessment visit. The ITT population was the primary sample and included: Pregabalin 165 mg: 100, Pregabalin 330 mg: 112, Placebo: 109.
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 98 | 111 | 109
percentage of participants
  Responder | 37.8 | 45.9 | 35.8
  Non-responder | 62.2 | 54.1 | 64.2
Statistical Analysis 1: Comparison: Pregabalin 165 mg vs Placebo; A 2-sided Cochran-Mantel-Haenszel test stratified by geographical region (U.S., Europe, Asia, or Rest of the World) was used to calculate the p-value. No adjustments for multiplicity were taken; Test type: Superiority; p = 0.752, Cochran-Mantel-Haenszel — Statistical testing was done at alpha = 0.05 level, two-sided
Statistical Analysis 2: Comparison: Pregabalin 330 mg vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.125, Cochran-Mantel-Haenszel — Statistical testing was done at alpha = 0.05 level, two-sided

3. Secondary Outcome: Percentage Change From Baseline in 28-day Partial Seizure Rate During the Double-blind Treatment Phase
Description: as for outcome 1
Time Frame: Week 0 to Week 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ln (seizures per 28 days)
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 98 | 111 | 109
ln (seizures per 28 days) | -15.00 (11.668) | -31.54 (10.772) | -5.70 (10.918)
Statistical Analysis 1: Comparison: Pregabalin 165 mg vs Placebo; ANCOVA model was used to calculate the p-value; Test type: Superiority; p = 0.5404, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided; LS Mean Difference = -9.30, 95% CI 2-sided [-39.16 to 20.56] — Value is percent reduction in seizures relative to placebo
Statistical Analysis 2: Comparison: Pregabalin 330 mg vs Placebo; ANCOVA model was used to calculate the p-value; Test type: Superiority; p = 0.0786, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided; LS Mean Difference = -25.84, 95% CI 2-sided [-54.64 to 2.97] — Value is percent reduction in seizures relative to placebo

4. Secondary Outcome: Frequency of Secondary Generalized Tonic-clonic Seizures (SGTC) During the Double-blind Treatment Phase
Description: Seizures were recorded and documented in a daily Seizure Diary by the participants, family member, caregiver, or legal guardian. Simple partial seizures without a visible motor component (ie, lacking visible movements during the seizure) were not counted toward eligibility, or in the primary or secondary efficacy analyses.
Time Frame: Week 0 to Week 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: seizures per 28 days
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 98 | 111 | 109
seizures per 28 days | 3.99 (8.667) | 4.43 (14.736) | 7.51 (24.979)
Statistical Analysis 1: Comparison: Pregabalin 165 mg vs Placebo; A generalized linear model accounting for treatment and geographical region as fixed effects and baseline seizure frequency as a covariate was used to calculate the p-value. This generalized linear model assumed that the SGTC seizure frequency was from a Poisson distribution with a canonical log link function; Test type: Superiority; p = 0.6073, Generalized linear model (GLM) — Statistical testing was done at alpha = 0.05 level, two-sided; LS Mean Difference = -0.11, 95% CI 2-sided [-0.53 to 0.31]
Statistical Analysis 2: Comparison: Pregabalin 330 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.4109, GLM — Statistical testing was done at alpha = 0.05 level, two-sided; LS Mean Difference = -0.16, 95% CI 2-sided [-0.53 to 0.22]

5. Secondary Outcome: Log Transformed 28-day SGTC Rate for All SGTCs During the Double-blind Maintenance Phase
Description: as for outcome 1
Time Frame: Week 2 to Week 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ln (seizures per 28 days)
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 96 | 110 | 109
ln (seizures per 28 days) | 0.46 (0.049) | 0.48 (0.045) | 0.48 (0.046)
Statistical Analysis 1: Comparison: Pregabalin 165 mg vs Placebo; ANCOVA model with the following fixed terms was used to calculate the p-value: loge (baseline 28-day seizure rate + 1) as a coninuous covariate, sites pooled by geographic region (ie, U.S., Europe, Asia, rest of the world), and treatment group (placebo, pregabalin 165 mg CR, pregabalin 330 mg CR); Test type: Superiority; p = 0.8268, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided; LS Mean Difference = -1.38, 95% CI 2-sided [-12.97 to 11.75] — Value is percent reduction in seizures relative to placebo
Statistical Analysis 2: Comparison: Pregabalin 330 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.9024, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided; LS Mean Difference = 0.75, 95% CI 2-sided [-10.69 to 13.66] — Value is percent reduction in seizures relative to placebo

6. Secondary Outcome: Percentage of Participants With ≥50% Reduction in 28-day SGTC Seizure Rate From Baseline During the Double-blind Treatment Phase
Description: as for outcome 4
Time Frame: Week 0 to Week 14
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 96 | 108 | 105
percentage of participants | 1.0 | 1.9 | 1.9
Statistical Analysis 1: Comparison: Pregabalin 165 mg vs Placebo; A 2-sided Cochran-Mantel-Haenszel test stratified by geographical region (U.S., Europe, Asia, or Rest of the World) wtih percentage of responders summarized by treatment group was used to calculate the p-value; Test type: Superiority; p = 0.670, Cochran-Mantel-Haenszel — Statistical testing was done at alpha = 0.05 level, two-sided
Statistical Analysis 2: Comparison: Pregabalin 330 mg vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.927, Cochran-Mantel-Haenszel — Statistical testing was done at alpha = 0.05 level, two-sided

7. Secondary Outcome: Loge 28-day Seizure Rate for All Partial Onset Seizures During the Double-blind Maintenance Phase
Description: as for outcome 1
Time Frame: Week 2 to Week 14
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ln(28-day seizure rate)
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 96 | 110 | 109
ln(28-day seizure rate) | 1.91 (0.070) | 1.77 (0.064) | 1.88 (0.065)
Statistical Analysis 1: Comparison: Pregabalin 165 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.8034, ANCOVA — Statistical testing was done at 95% confidence intervals, two-sided, least square means and their standard errors; LS Mean Difference = 2.28, 95% CI 2-sided [-14.37 to 22.15] — Value is percent reduction in seizures relative to placebo
Statistical Analysis 2: Comparison: Pregabalin 330 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.1905, ANCOVA — Statistical testing was done at 95% confidence intervals, two-sided, least square means and their standard errors; LS Mean Difference = -10.78, 95% CI 2-sided [-24.81 to 5.87] — Value is percent reduction in seizures relative to placebo

8. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale - Anxiety (HADS-A) Total Score at Week 14
Description: HADS: participant rated questionnaire with 2 subscales. HADS-A assesses state of generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks); HADS-D assesses state of lost interest and diminished pleasure response (lowering of hedonic tone). Each subscale comprised of 7 items with range 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Total score 0 to 21 for each subscale; higher score indicates greater severity of anxiety and depression symptoms.
Time Frame: Baseline, Week 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 93 | 103 | 101
units on a scale | -0.8 (3.34) | -0.4 (3.19) | -0.5 (3.13)
Statistical Analysis 1: Comparison: Pregabalin 165 mg vs Placebo; ANCOVA model with the following fixed terms was used to calculate the p-value: HADS-A baseline score as a coninuous covariate, sites pooled by geographic region (ie, U.S., Europe, Asia, rest of the world), and treatment group (placebo, pregabalin 165 mg controlled-release (CR), pregabalin 330 mg CR). No adjustments for multiplicity were taken; Test type: Superiority; p = 0.4650, ANCOVA — Statistical testing was done at 95% confidence intervals, two-sided, least square means and their standard errors; LS Mean Difference = -0.3, 95% CI 2-sided [-1.1 to 0.5]
Statistical Analysis 2: Comparison: Pregabalin 330 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.9692, ANCOVA — Statistical testing was done at 95% confidence intervals, two-sided, least square means and their standard errors; LS Mean Difference = 0.0, 95% CI 2-sided [-0.8 to 0.8]

9. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale - Depression (HADS-D) Total Score at Week 14
Description: as for outcome 8
Time Frame: Baseline, Week 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 93 | 103 | 101
units on a scale | -0.5 (3.16) | -0.8 (3.49) | -0.1 (3.17)
Statistical Analysis 1: Comparison: Pregabalin 165 mg vs Placebo; ANCOVA model with the following fixed terms was used to calculate the p-value: HADS-D baseline score as a coninuous covariate, sites pooled by geographic region (ie, U.S., Europe, Asia, rest of the world), and treatment group (placebo, pregabalin 165 mg controlled-release (CR), pregabalin 330 mg CR). No adjustments for multiplicity were taken; Test type: Superiority; p = 0.2693, ANCOVA — Statistical testing was done at 95% confidence intervals, two-sided, least square means and their standard errors; LS Mean Difference = -0.5, 95% CI 2-sided [-1.3 to 0.4]
Statistical Analysis 2: Comparison: Pregabalin 330 mg vs Placebo; [analysis description as in outcome 9, analysis 1]; Test type: Superiority; p = 0.1893, ANCOVA — Statistical testing was done at 95% confidence intervals, two-sided, least square means and their standard errors; LS Mean Difference = -0.5, 95% CI 2-sided [-1.4 to 0.3]

10. Secondary Outcome: Change From Baseline in Medical Outcomes Study Sleep Scale (MOS-SS) - Sleep Disturbance Score at Week 14
Description: Participant-rated 12-item questionnaire to assess key constructs of sleep over the past week. 7 subscales: sleep disturbance, snoring, awakened short of breath or with headache, sleep adequacy, and somnolence (range:0-100); sleep quantity (range:0-24), and optimal sleep (yes: 1, no: 0). 6 and 9 item index measures of sleep disturbance were constructed to provide composite scores. Scores are transformed (actual raw score minus lowest possible score divided by possible raw score range * 100); total score range: 0 to 100; higher score = greater intensity of attribute.
Time Frame: Baseline, Week 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 93 | 103 | 101
units on a scale | -3.9 (19.89) | -1.5 (17.93) | -1.9 (14.10)
Statistical Analysis 1: Comparison: Pregabalin 165 mg vs Placebo; ANCOVA model with the following fixed terms was used to calculate the p-value: sleep disturbance score at baseline as a coninuous covariate, sites pooled by geographic region (ie, U.S., Europe, Asia, rest of the world), and treatment group (placebo, pregabalin 165 mg CR, pregabalin 330 mg CR); Test type: Superiority; p = 0.7347, ANOVA — Statistical testing was done at alpha = 0.05 level, two-sided; LS Mean Difference = -0.8, 95% CI 2-sided [-5.2 to 3.6]
Statistical Analysis 2: Comparison: Pregabalin 330 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.8971, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided; LS Mean Difference = 0.3, 95% CI 2-sided [-4.0 to 4.6]

11. Secondary Outcome: Change From Baseline in MOS-SS - Snoring Score at Week 14
Description: as for outcome 10
Time Frame: Baseline, Week 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 92 | 103 | 101
units on a scale | -3.5 (25.44) | 5.4 (26.00) | -0.6 (22.71)
Statistical Analysis 1: Comparison: Pregabalin 165 mg vs Placebo; ANCOVA model with the following fixed terms was used to calculate the p-value: snoring score at baseline as a coninuous covariate, sites pooled by geographic region (ie, U.S., Europe, Asia, rest of the world), and treatment group (placebo, pregabalin 165 mg CR, pregabalin 330 mg CR); Test type: Superiority; p = 0.3972, ANOVA — Statistical testing was done at alpha = 0.05 level, two-sided; LS Mean Difference = -2.7, 95% CI 2-sided [-9.1 to 3.6]
Statistical Analysis 2: Comparison: Pregabalin 330 mg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.0319, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided; LS Mean Difference = 6.7, 95% CI 2-sided [0.6 to 12.9]

12. Secondary Outcome: Change From Baseline in MOS-SS - Awaken Short of Breath or With Headache Score at Week 14
Description: as for outcome 10
Time Frame: Baseline, Week 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 93 | 103 | 101
units on a scale | 0.2 (20.75) | 1.0 (24.48) | -0.8 (18.96)
Statistical Analysis 1: Comparison: Pregabalin 165 mg vs Placebo; ANCOVA model with the following fixed terms was used to calculate the p-value: awaken short of breath or with headache score at baseline as a coninuous covariate, sites pooled by geographic region (ie, U.S., Europe, Asia, rest of the world), and treatment group (placebo, pregabalin 165 mg CR, pregabalin 330 mg CR); Test type: Superiority; p = 0.7708, ANOVA — Statistical testing was done at alpha = 0.05 level, two-sided; LS Mean Difference = 0.8, 95% CI 2-sided [-4.4 to 5.9]
Statistical Analysis 2: Comparison: Pregabalin 330 mg vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.3560, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided; LS Mean Difference = 2.4, 95% CI 2-sided [-2.7 to 7.4]

13. Secondary Outcome: Change From Baseline in MOS-SS - Quantity of Sleep (Hours) at Week 14
Description: as for outcome 10
Time Frame: Baseline, Week 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 92 | 103 | 100
hours | 0.2 (1.31) | -0.1 (1.18) | -0.1 (1.25)
Statistical Analysis 1: Comparison: Pregabalin 165 mg vs Placebo; ANCOVA model with the following fixed terms was used to calculate the p-value: quantity of sleep at baseline as a coninuous covariate, sites pooled by geographic region (ie, U.S., Europe, Asia, rest of the world), and treatment group (placebo, pregabalin 165 mg CR, pregabalin 330 mg CR); Test type: Superiority; p = 0.1129, ANOVA — Statistical testing was done at alpha = 0.05 level, two-sided; LS Mean Difference = 0.2, 95% CI 2-sided [-0.1 to 0.5]
Statistical Analysis 2: Comparison: Pregabalin 330 mg vs Placebo; [analysis description as in outcome 13, analysis 1]; Test type: Superiority; p = 0.9388, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided; LS Mean Difference = 0.0, 95% CI 2-sided [-0.3 to 0.3]

14. Secondary Outcome: Change From Baseline in MOS-SS - Sleep Adequacy Score at Week 14
Description: as for outcome 10
Time Frame: Baseline, Week 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 93 | 103 | 101
units on a scale | 2.3 (31.14) | -1.7 (31.44) | -1.5 (24.55)
Statistical Analysis 1: Comparison: Pregabalin 165 mg vs Placebo; ANCOVA model with the following fixed terms was used to calculate the p-value: sleep adequacy score at baseline as a coninuous covariate, sites pooled by geographic region (ie, U.S., Europe, Asia, rest of the world), and treatment group (placebo, pregabalin 165 mg CR, pregabalin 330 mg CR); Test type: Superiority; p = 0.9053, ANOVA — Statistical testing was done at alpha = 0.05 level, two-sided; LS Mean Difference = -0.4, 95% CI 2-sided [-7.5 to 6.6]
Statistical Analysis 2: Comparison: Pregabalin 330 mg vs Placebo; [analysis description as in outcome 14, analysis 1]; Test type: Superiority; p = 0.6371, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided; LS Mean Difference = -1.6, 95% CI 2-sided [-8.5 to 5.2]

15. Secondary Outcome: Change From Baseline in MOS-SS - Sleep Somnolence Score at Week 14
Description: as for outcome 10
Time Frame: Baseline, Week 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 93 | 103 | 101
units on a scale | -0.5 (17.29) | 5.2 (19.42) | 5.0 (18.72)
Statistical Analysis 1: Comparison: Pregabalin 165 mg vs Placebo; ANCOVA model with the following fixed terms was used to calculate the p-value: sleep somnolence score at baseline as a coninuous covariate, sites pooled by geographic region (ie, U.S., Europe, Asia, rest of the world), and treatment group (placebo, pregabalin 165 mg CR, pregabalin 330 mg CR); Test type: Superiority; p = 0.0119, ANOVA — Statistical testing was done at alpha = 0.05 level, two-sided; LS Mean Difference = -6.4, 95% CI 2-sided [-11.4 to -1.4]
Statistical Analysis 2: Comparison: Pregabalin 330 mg vs Placebo; [analysis description as in outcome 15, analysis 1]; Test type: Superiority; p = 0.9909, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided; LS Mean Difference = 0.0, 95% CI 2-sided [-4.9 to 4.8]

16. Secondary Outcome: Change From Baseline in MOS-SS - Sleep Problems Index I Score at Week 14
Description: as for outcome 10
Time Frame: Baseline, Week 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 93 | 103 | 101
units on a scale | -2.2 (16.91) | 0.4 (16.43) | 0.3 (12.62)
Statistical Analysis 1: Comparison: Pregabalin 165 mg vs Placebo; ANCOVA model with the following fixed terms was used to calculate the p-value: sleep problems index I score at baseline as a coninuous covariate, sites pooled by geographic region (ie, U.S., Europe, Asia, rest of the world), and treatment group (placebo, pregabalin 165 mg CR, pregabalin 330 mg CR); Test type: Superiority; p = 0.5903, ANOVA — Statistical testing was done at alpha = 0.05 level, two-sided; LS Mean Difference = -1.1, 95% CI 2-sided [-5.0 to 2.8]
Statistical Analysis 2: Comparison: Pregabalin 330 mg vs Placebo; [analysis description as in outcome 16, analysis 1]; Test type: Superiority; p = 0.7126, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided; LS Mean Difference = 0.7, 95% CI 2-sided [-3.1 to 4.5]

17. Secondary Outcome: Change From Baseline in Medical Outcomes Study Sleep Scale (MOS-SS) - Sleep Problems Index II Score at Week 14
Description: as for outcome 10
Time Frame: Baseline, Week 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 93 | 103 | 101
units on a scale | -2.4 (15.62) | 0.7 (14.53) | 0.7 (11.30)
Statistical Analysis 1: Comparison: Pregabalin 165 mg vs Placebo; ANCOVA model with the following fixed terms was used to calculate the p-value: sleep problems index II score at baseline as a coninuous covariate, sites pooled by geographic region (ie, U.S., Europe, Asia, rest of the world), and treatment group (placebo, pregabalin 165 mg CR, pregabalin 330 mg CR); Test type: Superiority; p = 0.2431, ANOVA — Statistical testing was done at alpha = 0.05 level, two-sided; LS Mean Difference = -2.1, 95% CI 2-sided [-5.8 to 1.5]
Statistical Analysis 2: Comparison: Pregabalin 330 mg vs Placebo; [analysis description as in outcome 17, analysis 1]; Test type: Superiority; p = 0.8654, ANCOVA — Statistical testing was done at alpha = 0.05 level, two-sided; LS Mean Difference = 0.3, 95% CI 2-sided [-3.2 to 3.8]

18. Secondary Outcome: Percent of Participants Reporting Optimal Sleep on the MOS-SS - Optimal Sleep Subscale
Description: Optimal sleep was considered between 7 to 8 hours of average sleep per night inclusive, while average sleep less than or greater than the 7 to 8 hour of average sleep per night was non-optimal.
Time Frame: Week 14
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 93 | 103 | 103
percentage of participants | 67.7 | 60.2 | 60.2
Statistical Analysis 1: Comparison: Pregabalin 165 mg vs Placebo; Logistic regression model was used to calculate the p-value, with the fixed effects for sites pooled by geographic region (ie, U.S., Europe, Asia, rest of the world), and treatment group (placebo, pregabalin 165 mg controlled-release (CR), pregabalin 330 mg CR), average hours per night of sleep at baseline as a coninuous covariate, and optimal sleep at Week 14 as dependent variable. No adjustments for multiplicity were taken; Test type: Superiority; p = 0.3241, Regression, Logistic — Statistical testing was done at alpha = 0.05 level, two-sided; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.74 to 2.50]
Statistical Analysis 2: Comparison: Pregabalin 330 mg vs Placebo; [analysis description as in outcome 18, analysis 1]; Test type: Superiority; p = 0.8932, Regression, Logistic — Statistical testing was done at alpha = 0.05 level, two-sided; Odds Ratio (OR) = 0.96, 95% CI 2-sided [0.54 to 1.71]

19. Secondary Outcome: Benefit, Satisfaction, and Willingness to Continue Measure (BSW): Benefit From Treatment Question
Description: The BSW consisted of 3 single-item measures designed to capture the participant's perception of the effect of treatment in terms of the relative benefit, their satisfaction, and their intention or willingness to continue on therapy. The BSW was read aloud to the participant by the investigator or designated center personnel and then was given to the participant to complete independently.
Time Frame: Week 14
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 100 | 112 | 109
percentage of participants
  No | 12.0 | 17.9 | 22.0
  Little benefit | 31.0 | 23.2 | 33.0
  Much benefit | 54.0 | 56.3 | 42.2
  Not done | 2.0 | 1.8 | 1.8
  Missing | 1.0 | 0.9 | 0.9

20. Secondary Outcome: BSW: Satisfaction From Treatment Question
Description: as for outcome 19
Time Frame: Week 14
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 100 | 112 | 109
percentage of participants
  No | 13.0 | 17.9 | 23.9
  Yes | 84.0 | 80.4 | 73.4
  Missing | 3.0 | 1.8 | 2.8

21. Secondary Outcome: BSW: Willingness to Continue Question
Description: as for outcome 19
Time Frame: Week 14
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 100 | 112 | 109
percentage of participants
  No | 18.0 | 22.3 | 26.6
  Yes | 79.0 | 75.9 | 70.6
  Missing | 3.0 | 1.8 | 2.8

22. Secondary Outcome: Percentage of Participants With New or Intensified Physical Examination Findings During the Double-blind Treatment Phase
Description: Physical examinations included general appearance (including hight at baseline), vital sign (sitting heart rate and sitting blood pressure), weight, skin (examination for the presence of rash), HEENT (examinatin of head, eyes, ears, nose and throat), chest ausculation of lung fields), cardiovascular (ausculatin of heart sounds (S1 and S2) and for the presence of murmurs, gallops, or rubs), gastrointestinal (abdominal rigidity and tenderness), an extremities (e.g. edema). Clinically significant physical examination abnormalities were considered as adverse events based on investigator's discretion.
Time Frame: Day 1 to Week 15
Population: The safety population included all randomized participants who took at least one dose of the study medication. The safety population consisted of: Pregabalin 165 mg: 100, Pregabalin 330 mg: 113, Placebo: 110.
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 100 | 113 | 110
percentage of participants
  General | 1.0 | 2.7 | 0.0
  Skin | 2.0 | 6.2 | 4.5
  Head | 1.0 | 1.8 | 0.0
  Ears | 3.0 | 1.8 | 0.9
  Eyes | 1.0 | 2.7 | 3.6
  Nose | 0.0 | 0.0 | 1.8
  Throat | 0.0 | 0.0 | 1.8
  Lungs | 0.0 | 0.0 | 0.0
  Heart | 1.0 | 0.0 | 0.0
  Abdomen | 0.0 | 0.0 | 0.0
  Extremities | 2.0 | 2.7 | 1.8
  Other | 14.0 | 7.1 | 10.9

23. Secondary Outcome: Percentage of Participants With New or Intensified Neurological Examination Findings During the Double-blind Treatment Phase
Description: Neurological examinations included level of consciousness, mental status, cranial nerve assessment, muscle strength, reflexes, pin prick and vibratory sensation (the latter using a 128-Hz tuning fork), coordination and gait.
Time Frame: Day 1 to Week 15
Population: as for outcome 22
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 100 | 113 | 110
percentage of participants
  None | 79.0 | 78.8 | 68.2
  Any | 21.0 | 21.2 | 31.8
  Coordination | 1.0 | 1.8 | 1.8
  Cranial nerve function: number analyzed (Participants) | 99 | 111 | 108
  Cranial nerve function | 0.0 | 0.9 | 0.0
  Cranial nerve II: number analyzed (Participants) | 99 | 111 | 108
  Cranial nerve II | 0.0 | 0.0 | 0.0
  Cranial nerve III | 0.0 | 0.0 | 1.8
  Cranial nerve V: number analyzed (Participants) | 99 | 111 | 108
  Cranial nerve V | 0.0 | 0.0 | 0.0
  Cranial nerve VII: number analyzed (Participants) | 99 | 111 | 108
  Cranial nerve VII | 1.0 | 0.0 | 0.9
  Cranial nerve VIII: number analyzed (Participants) | 99 | 111 | 108
  Cranial nerve VIII | 0.0 | 0.9 | 0.0
  Cranial nerve XI: number analyzed (Participants) | 99 | 111 | 108
  Cranial nerve XI | 0.0 | 0.0 | 0.0
  Deep tendon reflexes | 3.0 | 1.8 | 2.7
  Gait and station | 0.0 | 0.0 | 0.9
  Level of consciousness | 0.0 | 0.0 | 0.9
  Mental state | 1.0 | 1.8 | 1.8
  Motor function | 1.0 | 2.7 | 3.6
  Muscle strength: number analyzed (Participants) | 99 | 111 | 108
  Muscle strength | 2.0 | 0.0 | 1.9
  Pain sensation: number analyzed (Participants) | 99 | 111 | 108
  Pain sensation | 0.0 | 0.0 | 1.9
  Reflexes: number analyzed (Participants) | 99 | 111 | 108
  Reflexes | 1.0 | 0.9 | 1.9
  Vibration: number analyzed (Participants) | 99 | 111 | 108
  Vibration | 11.1 | 10.8 | 12.0

24. Secondary Outcome: Percentage of Participants With Self-injurious or Suicidal Ideation or Behavior on Columbia Classification Algorithm of Suicide Assessment (C-CASA)
Description: C-CASA is described as a standardized suicidal rating system. The C-CASA has eight categories (4 suicidal events: completed suicide, suicide attempt, preparatory act toward imminent suicidal behavior (PAISB), and suicidal ideation; 2 nonsuicidal events: self-injurious behavior, no suicidal intent (SIB-NSI) and other no deliberate self-harm, and 2 indeterminate or potentially suicidal events: self-injurious behavior, suicidal intent unknown and not enough information) that distinguish suicidal events from nonsuicidal events and indeterminate or potentially suicidal events.
Time Frame: Week -8 (Screening), Week 0 (Baseline), and Week 14 (double-blind treatment phase)
Population: as for outcome 22
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 100 | 113 | 110
percentage of participants
  Suicide attempt (Lifetime prior to Screening) | 2.0 | 1.8 | 5.5
  PAISB (Lifetime prior to Screening) | 1.0 | 1.8 | 4.5
  Suicidal ideation (Lifetime prior to Screening) | 11.0 | 10.6 | 14.5
  SIB-NSI (Lifetime prior to Screening) | 1.0 | 0.9 | 0.9
  Suicide attempts at Week 0 | 1.0 | 0.9 | 0.0
  PAISB at Week 0 | 0.0 | 0.9 | 0.0
  Suicidal ideation at Week 0 | 8.0 | 7.1 | 2.7
  SIB-NSI at Week 0 | 1.0 | 0.0 | 0.0
  Suicidal ideation at Week 14 | 4.0 | 2.7 | 1.8

25. Secondary Outcome: Percentage of Participants With a Relevant Increase in Sitting Blood Pressure (BP) From Baseline During the Double-blind Treatment Phase
Description: Physical examinations included general appearance (including hight at baseline), vital sign (sitting heart rate and sitting blood pressure), weight, skin (examination for the presence of rash), HEENT (examinatin of head, eyes, ears, nose and throat), chest (ausculation of lung fields), cardiovascular (ausculatin of heart sounds (S1 and S2) and for the presence of murmurs, gallops, or rubs), gastrointestinal(abdominal rigidity and tenderness), an extremities (e.g. edema).
Time Frame: Day 1 to Week 15
Population: as for outcome 22
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 99 | 110 | 108
percentage of participants
  Maximum increase in systolic BP ≥30 mmHg | 1.0 | 1.8 | 0.9
  Maximum increase in diastolic BP ≥20 mmHg | 5.1 | 5.5 | 2.8

26. Secondary Outcome: Percentage of Participants With Corrected QT (QTc) Interval Greater Than or Equal to 450 ms
Description: The original ECG was reviewed by the investigator and kept on site as part of source documentation. A central ECG reader was also used for this study. QT interval corrected using the Fridericia formula (QTcF) and QT interval corrected using the Bazett's formula (QTcB) were calculated.
Time Frame: Week 15
Population: as for outcome 22
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 100 | 113 | 110
percentage of participants
  Maximum QTcB 450 - <480 | 8.0 | 5.3 | 10.0
  Maximum QTcB 480 - <500 | 1.0 | 0.0 | 0.9
  Maximum QTcB ≥500 | 0.0 | 1.8 | 0.0
  Maximum QTcF 450 - <480 | 3.0 | 2.7 | 3.6
  Maximum QTcF 480 - <500 | 1.0 | 0.0 | 0.0
  Maximum QTcF ≥500 | 0.0 | 0.0 | 0.0

27. Secondary Outcome: Percentage of Participants With Relevant ECG Interval-increases From Baseline During the Double-blind Treatment Phase
Description: The original ECG was reviewed by the investigator and kept on site as part of source documentation. A central ECG reader was also used for this study. 25/50% represents ≥25% or ≥50% increase over baseline respectively, based on cut points. Cut points are 100 ms for QRS and 200 ms for PR.
Time Frame: Week 15
Population: as for outcome 22
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 100 | 113 | 110
percentage of participants
  Max PR interval rise:%change≥25/50%: number analyzed (Participants) | 92 | 104 | 96
  Max PR interval rise:%change≥25/50% | 1.1 | 1.0 | 2.1
  Max QRS complex rise:%change≥25/50%: number analyzed (Participants) | 92 | 104 | 96
  Max QRS complex rise:%change≥25/50% | 1.1 | 1.9 | 1.0
  Max. QTcB interval rise: 30≤x<60: number analyzed (Participants) | 93 | 104 | 97
  Max. QTcB interval rise: 30≤x<60 | 5.4 | 1.9 | 3.1
  Max. QTcB interval rise: ≥60: number analyzed (Participants) | 93 | 104 | 97
  Max. QTcB interval rise: ≥60 | 0.0 | 1.9 | 0.0
  Max. QTcF interval rise: 30≤x<60: number analyzed (Participants) | 93 | 104 | 97
  Max. QTcF interval rise: 30≤x<60 | 3.2 | 1.9 | 2.1
  Max. QTcF interval rise: ≥60: number analyzed (Participants) | 93 | 104 | 97
  Max. QTcF interval rise: ≥60 | 0.0 | 0.0 | 0.0

28. Secondary Outcome: Percentage of Participants With Laboratory Test Abnormalities During the Study
Description: Laboratory samples in hematology, chemistry, and urinalysis were analyzed by a cental laboratory. Any laboratory value that was identified as clinically significant was reported as an AE. LLN: Lower limit of normal, ULN: Uper limit of normal, RBC: Red Blood Cell, WBC: White Blood Cell, AST: Aspartate Aminotransferase, ALT: Alanine Aminotransferase, BUN: Blood Urea Nitrogen
Time Frame: Day 1 to Week 15
Population: as for outcome 22
Measure: Number; unit: percentage of participants
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Number analyzed (Participants) | 99 | 111 | 108
percentage of participants
  Hemoglobin (HGB) <0.8xLLN ,: number analyzed (Participants) | 98 | 109 | 107
  Hemoglobin (HGB) <0.8xLLN , | 1.0 | 0.9 | 0.9
  Hematocrit (HCT) <0.8xLLN: number analyzed (Participants) | 96 | 107 | 107
  Hematocrit (HCT) <0.8xLLN | 0.0 | 0.9 | 0.0
  RBC Count <0.8xLLN: number analyzed (Participants) | 98 | 109 | 107
  RBC Count <0.8xLLN | 0.0 | 0.0 | 0.0
  Platelets <0.5xLLN: number analyzed (Participants) | 95 | 108 | 105
  Platelets <0.5xLLN | 0.0 | 0.0 | 0.0
  Platelets >1.75xULN: number analyzed (Participants) | 95 | 108 | 105
  Platelets >1.75xULN | 0.0 | 0.0 | 0.0
  WBC Count <0.6xLLN: number analyzed (Participants) | 98 | 109 | 107
  WBC Count <0.6xLLN | 0.0 | 0.9 | 0.0
  White Blood Cell Count >1.5xULN: number analyzed (Participants) | 98 | 109 | 107
  White Blood Cell Count >1.5xULN | 0.0 | 0.0 | 0.0
  Lymphocytes (absolute) <0.8xLLN: number analyzed (Participants) | 96 | 109 | 106
  Lymphocytes (absolute) <0.8xLLN | 4.2 | 0.9 | 1.9
  Lymphocytes (absolute) >1.2xULN: number analyzed (Participants) | 96 | 109 | 106
  Lymphocytes (absolute) >1.2xULN | 2.1 | 1.8 | 3.8
  Lymphocytes (%) <0.8xLLN: number analyzed (Participants) | 96 | 109 | 106
  Lymphocytes (%) <0.8xLLN | 0.0 | 0.0 | 1.9
  Lymphocytes (%) >1.2xULN: number analyzed (Participants) | 96 | 109 | 106
  Lymphocytes (%) >1.2xULN | 1.0 | 0.0 | 0.9
  Neutrophils (absolute) <0.8xLLN: number analyzed (Participants) | 96 | 109 | 106
  Neutrophils (absolute) <0.8xLLN | 3.1 | 1.8 | 1.9
  Neutrophils (absolute) >1.2xULN: number analyzed (Participants) | 96 | 109 | 106
  Neutrophils (absolute) >1.2xULN | 0.0 | 0.0 | 1.9
  Neutrophils (%) <0.8xLLN: number analyzed (Participants) | 96 | 109 | 106
  Neutrophils (%) <0.8xLLN | 1.0 | 0.0 | 0.0
  Neutrophils (%) >1.2xULN: number analyzed (Participants) | 96 | 109 | 106
  Neutrophils (%) >1.2xULN | 0.0 | 0.0 | 0.0
  Basophils (absolute) >1.2xULN: number analyzed (Participants) | 96 | 109 | 106
  Basophils (absolute) >1.2xULN | 0.0 | 0.0 | 0.0
  Basophils (%) >1.2xULN: number analyzed (Participants) | 96 | 109 | 106
  Basophils (%) >1.2xULN | 0.0 | 0.0 | 0.0
  Eosinophils (absolute) >1.2xULN: number analyzed (Participants) | 96 | 109 | 106
  Eosinophils (absolute) >1.2xULN | 3.1 | 3.7 | 1.9
  Eosinophils (%) >1.2xULN: number analyzed (Participants) | 96 | 109 | 106
  Eosinophils (%) >1.2xULN | 6.3 | 4.6 | 3.8
  Monocytes (absolute) >1.2xULN: number analyzed (Participants) | 96 | 109 | 106
  Monocytes (absolute) >1.2xULN | 0.0 | 1.8 | 0.0
  Monocytes (%) >1.2xULN: number analyzed (Participants) | 96 | 109 | 106
  Monocytes (%) >1.2xULN | 1.0 | 0.0 | 0.0
  Total Bilirubin >1.5xULN: number analyzed (Participants) | 98 | 111 | 107
  Total Bilirubin >1.5xULN | 0.0 | 0.0 | 0.0
  AST >3.0xULN: number analyzed (Participants) | 98 | 111 | 107
  AST >3.0xULN | 0.0 | 0.0 | 0.0
  ALT >3.0xULN: number analyzed (Participants) | 98 | 111 | 107
  ALT >3.0xULN | 0.0 | 0.0 | 0.0
  Alkaline Phosphatase >3.0xULN: number analyzed (Participants) | 98 | 111 | 107
  Alkaline Phosphatase >3.0xULN | 0.0 | 0.0 | 0.0
  Total Protein <0.8xLLN: number analyzed (Participants) | 98 | 111 | 107
  Total Protein <0.8xLLN | 0.0 | 0.0 | 0.0
  Total Protein >1.2xULN: number analyzed (Participants) | 98 | 111 | 107
  Total Protein >1.2xULN | 0.0 | 0.0 | 0.0
  Albumin <0.8xLLN: number analyzed (Participants) | 98 | 111 | 107
  Albumin <0.8xLLN | 0.0 | 0.0 | 0.0
  Albumin >1.2xULN: number analyzed (Participants) | 98 | 111 | 107
  Albumin >1.2xULN | 0.0 | 0.0 | 0.0
  BUN >1.3xULN: number analyzed (Participants) | 98 | 111 | 107
  BUN >1.3xULN | 0.0 | 0.0 | 0.0
  Creatinine >1.3xULN: number analyzed (Participants) | 98 | 111 | 107
  Creatinine >1.3xULN | 0.0 | 0.0 | 0.0
  Uric Acid >1.2xULN: number analyzed (Participants) | 98 | 111 | 107
  Uric Acid >1.2xULN | 1.0 | 0.9 | 0.0
  Sodium <0.95xLLN: number analyzed (Participants) | 97 | 111 | 106
  Sodium <0.95xLLN | 1.0 | 0.0 | 0.0
  Sodium >1.05xULN: number analyzed (Participants) | 97 | 111 | 106
  Sodium >1.05xULN | 0.0 | 0.0 | 0.0
  Potassium <0.9xLLN: number analyzed (Participants) | 98 | 111 | 107
  Potassium <0.9xLLN | 2.0 | 0.0 | 0.0
  Potassium >1.1xULN: number analyzed (Participants) | 98 | 111 | 107
  Potassium >1.1xULN | 1.0 | 0.0 | 0.0
  Chloride <0.9xLLN: number analyzed (Participants) | 98 | 111 | 107
  Chloride <0.9xLLN | 0.0 | 0.0 | 0.0
  Chloride >1.1xULN: number analyzed (Participants) | 98 | 111 | 107
  Chloride >1.1xULN | 0.0 | 0.0 | 0.0
  Calcium <0.9xLLN: number analyzed (Participants) | 98 | 111 | 107
  Calcium <0.9xLLN | 0.0 | 0.0 | 0.0
  Calcium >1.1xULN: number analyzed (Participants) | 98 | 111 | 107
  Calcium >1.1xULN | 0.0 | 0.0 | 0.0
  Glucose <0.6xLLN: number analyzed (Participants) | 98 | 111 | 107
  Glucose <0.6xLLN | 0.0 | 0.0 | 0.0
  Glucose >1.5xULN: number analyzed (Participants) | 98 | 111 | 107
  Glucose >1.5xULN | 0.0 | 0.9 | 0.0
  Urine Specific Gravity <1.003: number analyzed (Participants) | 92 | 104 | 104
  Urine Specific Gravity <1.003 | 0.0 | 1.9 | 1.0
  Urine Specific Gravity >1.030: number analyzed (Participants) | 92 | 104 | 104
  Urine Specific Gravity >1.030 | 1.1 | 1.9 | 4.8
  Urine pH <4.5: number analyzed (Participants) | 93 | 105 | 104
  Urine pH <4.5 | 0.0 | 0.0 | 0.0
  Urine pH >8: number analyzed (Participants) | 93 | 105 | 104
  Urine pH >8 | 1.1 | 1.9 | 1.9
  Urine Glucose (qualitative) ≥1: number analyzed (Participants) | 94 | 106 | 105
  Urine Glucose (qualitative) ≥1 | 0.0 | 0.9 | 0.0
  Urine Ketones (qualitative) ≥1: number analyzed (Participants) | 94 | 106 | 105
  Urine Ketones (qualitative) ≥1 | 2.1 | 1.9 | 1.9
  Urine Protein (qualitative) ≥1: number analyzed (Participants) | 94 | 106 | 105
  Urine Protein (qualitative) ≥1 | 3.2 | 2.8 | 1.0
  Urine Blood/Hgb (qualitative) ≥1: number analyzed (Participants) | 94 | 106 | 105
  Urine Blood/Hgb (qualitative) ≥1 | 8.5 | 9.4 | 9.5
  Urine Nitrite ≥1: number analyzed (Participants) | 94 | 105 | 105
  Urine Nitrite ≥1 | 11.7 | 5.7 | 13.3
  Urine RBC ≥20: number analyzed (Participants) | 15 | 26 | 21
  Urine RBC ≥20 | 13.3 | 0.0 | 9.5
  Urine WBC ≥20: number analyzed (Participants) | 21 | 27 | 27
  Urine WBC ≥20 | 4.8 | 3.7 | 29.6

ADVERSE EVENTS:
Time Frame: From the time the participant provided informed consent, which was obtained prior to the participant's participation in the study, through and including 28 calendar days after the last administration of the investigational product.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one particpant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin 165 mg | Pregabalin 330 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 5/100 | 5/113 | 2/110
Other Adverse Events (participants affected / at risk) | 14/100 | 21/113 | 3/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin 165 mg (N=100) | Pregabalin 330 mg (N=113) | Placebo (N=110)
Bronchitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1 | 0
Complex partial seizures (Nervous system disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 1 | 1
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Hallucination (Psychiatric disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin 165 mg (N=100) | Pregabalin 330 mg (N=113) | Placebo (N=110)
Dizziness (Nervous system disorders) | 11 | 11 | 2
Fatigue (General disorders) | 3 | 6 | 1
Weight increased (Investigations) | 1 | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.